CLINICAL TRIAL: NCT07350876
Title: Promotion of a Standardized Diagnostic and Treatment Pathway for Polycystic Ovary Syndrome in Primary Care Based on a Bidirectional Referral System
Brief Title: Promotion of a Standardized Diagnostic and Treatment Pathway for Polycystic Ovary Syndrome Based on a Bidirectional Referral System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: [2022]214-002
Record Dates: First submitted 2025-12-30; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Polycystic Ovary Syndrome (PCOS)
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standardized PCOS Care + Lifestyle Intervention + Prebiotics (Experimental)
  Interventions: Dietary Supplement: Standardized Diagnostic and Treatment Pathways for PCOS + Lifestyle Intervention + Prebiotic Supplementation
- Standardized PCOS Care + Lifestyle Intervention (Active Comparator)
  Interventions: Behavioral: Standardized Diagnostic and Treatment Pathways for PCOS + Lifestyle Intervention

INTERVENTIONS:
Dietary Supplement: Standardized Diagnostic and Treatment Pathways for PCOS + Lifestyle Intervention + Prebiotic Supplementation — Participants will first undergo the same 12-week run-in phase as the control arm, during which standardized diagnostic and treatment pathways for PCOS combined with lifestyle intervention will be implemented uniformly. After completion of the run-in phase and randomization at Week 12, participants in the intervention arm will continue to receive lifestyle intervention and will additionally receive prebiotic supplementation for 8 weeks.
  Arms: Standardized PCOS Care + Lifestyle Intervention + Prebiotics
Behavioral: Standardized Diagnostic and Treatment Pathways for PCOS + Lifestyle Intervention — Participants will first undergo a 12-week run-in phase, during which standardized diagnostic and treatment pathways for PCOS combined with lifestyle intervention will be implemented uniformly. After completion of the run-in phase and randomization at Week 12, participants in the control arm will continue to receive lifestyle intervention alone for an additional 8 weeks.
  Arms: Standardized PCOS Care + Lifestyle Intervention

SUMMARY:
The goal of this clinical trial is to:

1. promote and optimize standardized diagnostic and treatment pathways for polycystic ovary syndrome (PCOS) and to investigate the clinical phenotypic characteristics of PCOS;
2. establish a bidirectional referral system and standardized referral pathways for PCOS;
3. comprehensively evaluate the effectiveness of standardized PCOS care pathways based on a bidirectional referral system;
4. collaborate with technical partners to develop an information-based clinical management platform for PCOS suitable for use in primary healthcare settings; and
5. investigate the effects of combined lifestyle intervention and prebiotic supplementation on insulin resistance and glucose-lipid metabolism in patients with PCOS.

The main questions this study aims to answer are:

1. What are the clinical phenotypic characteristics of PCOS, and how effective are standardized diagnostic and treatment pathways for PCOS?
2. What are the effects of combined lifestyle intervention and prebiotic supplementation, implemented within standardized diagnostic and treatment pathways for PCOS, on insulin resistance and glucose-lipid metabolism in patients with PCOS?

Researchers will compare standardized diagnostic and treatment pathways for PCOS before and after implementation to assess improvements in clinical outcomes in patients with PCOS, and will also compare lifestyle intervention with and without prebiotic supplementation to determine whether prebiotic supplementation can improve insulin resistance and glucos-lipid metabolism in patients with PCOS.

All participants will first undergo a 12-week run-in phase, during which standardized diagnostic and treatment pathways for PCOS combined with lifestyle intervention will be implemented uniformly. After completion of the run-in phase and randomization at Week 12, participants will be assigned to one of two parallel intervention arms. Participants in the control arm will continue to receive lifestyle intervention alone for an additional 8 weeks, without additional prebiotic supplementation. Participants in the intervention arm will continue to receive lifestyle intervention and will additionally receive prebiotic supplementation for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Female participants aged 18-50 years.
2. A diagnosis of PCOS based on the 2003 Rotterdam consensus, meeting at least two of the following three criteria: (i) oligo-ovulation and/or anovulation;(ii) clinical and/or biochemical signs of hyperandrogenism; or(iii) polycystic ovarian morphology on ultrasonography, defined as the presence of ≥12 follicles measuring 2-9 mm in diameter in each ovary and/or an ovarian volume ≥10 cm³.

Exclusion Criteria:

1. Patients with other serious medical conditions, including coronary heart disease (e.g., angina pectoris, myocardial infarction, history of coronary revascularization, or abnormal Q waves on electrocardiography), stroke (ischemic or hemorrhagic, including transient ischemic attack), or severe hepatic or renal dysfunction.
2. Patients with eating disorders or severe gastrointestinal diseases that may affect nutritional intervention outcomes.
3. Patients with any other medical condition associated with an estimated life expectancy of less than 5 years.
4. Patients with drug abuse, chronic alcoholism, alcohol dependence, or other addictive tendencies.
5. Patients who are unable to comply with dietary modification or lifestyle intervention or who are unlikely to adhere to follow-up visits.
6. Pregnant or lactating women, or those who have used oral contraceptives or glucagon-like peptide-1 (GLP-1) receptor agonists within the past 3 months.
7. Patients with a known allergy to prebiotics, those who have taken probiotics, prebiotics, or synbiotic supplements within the past 3 months, or those who have used antibiotics within the past 1 month.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 227 (Actual)
Dates: Start 2024-10-18 (Actual); Primary Completion 2025-12-13 (Actual); Study Completion 2025-12-13 (Actual)

PRIMARY OUTCOMES:
Clinical phenotypic characteristics of PCOS assessed by clinical evaluation | Baseline, Week 12, and Week 20
  1. Improvement in PCOS clinical phenotypes based on the Rotterdam criteria Improvement in PCOS clinical phenotypes will be assessed by trained study investigators based on changes in clinical manifestations, including menstrual cycle regularity, clinical hyperandrogenism, and gynecological ultrasound findings. Overall improvement will be evaluated based on changes in phenotype-specific clinical characteristics according to the Rotterdam criteria.
  2. Improvement in obesity-related metabolic phenotypes Improvement in obesity-related metabolic phenotypes will be assessed by trained study investigators based on changes in body weight status and metabolic health. Metabolic abnormality is defined as the presence of hypertension, impaired glucose metabolism, or dyslipidemia. Overall improvement will be evaluated based on changes in phenotype-specific characteristics related to body weight status and metabolic health.
Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) | Baseline, Week 12, and Week 20
  Insulin resistance will be assessed using the HOMA-IR, calculated from fasting plasma glucose and fasting insulin levels measured at predefined study time points. Outcomes will include HOMA-IR values reported as continuous variables and comparisons of changes in HOMA-IR between baseline and post-intervention time points and/or between intervention groups.

SECONDARY OUTCOMES:
Weight | Baseline, Week 12, and Week 20
Body Mass Index | Baseline, Week 12, and Week 20
Menstrual cycle regularity assessed by menstrual cycle length and frequency | Baseline, Week 12, and Week 20
  Menstrual cycle regularity will be assessed by the study investigators based on menstrual cycle length and cycle frequency, obtained from patient-reported menstrual history during study visits. Menstrual irregularity is defined as a menstrual cycle length <21 or >35 days, or fewer than 8 menstrual cycles per year.
Waist circumference | Baseline, Week 12, and Week 20
Waist-to-hip ratio | Baseline, Week 12, and Week 20
Blood pressure | Baseline, Week 12, and Week 20
Fasting plasma glucose | Baseline, Week 12, and Week 20
Fasting insulin | Baseline, Week 12, and Week 20
Triglycerides | Baseline, Week 12, and Week 20
Total cholesterol | Baseline, Week 12, and Week 20
Low-density lipoprotein cholesterol | Baseline, Week 12, and Week 20
High-density lipoprotein cholesterol | Baseline, Week 12, and Week 20
Uric acid | Baseline, Week 12, and Week 20

OTHER OUTCOMES:
Serum estradiol (E2) concentration | Baseline, Week 12, and Week 20
  Serum E2 concentrations will be measured in fasting serum samples collected at predefined study time points using standardized laboratory procedures. Outcomes will be reported as continuous variables, and changes in estradiol concentrations will be compared between baseline and post-intervention time points and/or between intervention groups.
Serum progesterone concentration | Baseline, Week 12, and Week 20
  Serum progesterone concentrations will be measured in fasting serum samples collected at predefined study time points using standardized laboratory procedures. Outcomes will be reported as continuous variables, and changes in progesterone concentrations will be compared between baseline and post-intervention time points and/or between intervention groups.
Serum total testosterone (TT) concentration | Baseline, Week 12, and Week 20
  Serum TT concentrations will be measured in fasting serum samples collected at predefined study time points using standardized laboratory procedures. Outcomes will be reported as continuous variables, and changes in total testosterone concentrations will be compared between baseline and post-intervention time points and/or between intervention groups.
Serum luteinizing hormone (LH) concentration | Baseline, Week 12, and Week 20
  LH concentrations will be measured in fasting serum samples collected at predefined study time points using standardized laboratory procedures. Outcomes will be reported as continuous variables, and changes in LH concentrations will be compared between baseline and post-intervention time points and/or between intervention groups.
Serum follicle-stimulating hormone (FSH) concentration | Baseline, Week 12, and Week 20
  Serum FSH concentrations will be measured in fasting serum samples collected at predefined study time points using standardized laboratory procedures. Outcomes will be reported as continuous variables, and changes in FSH concentrations will be compared between baseline and post-intervention time points and/or between intervention groups.
Serum anti-Müllerian hormone (AMH) concentration | Baseline, Week 12, and Week 20
  Serum anti-Müllerian hormone (AMH) concentrations will be measured in fasting serum samples collected at predefined study time points using standardized laboratory procedures. This outcome will be evaluated by trained study investigators.
Gut microbiota composition assessed by 16S rRNA gene sequencing | Baseline and Week 20
  Gut microbiota profiling will be conducted on fecal samples collected at predefined study time points using 16S rRNA gene sequencing. Outcomes will include measures of gut microbial diversity, relative abundances of bacterial taxa, and the identification of taxa showing significant changes between baseline and post-intervention time points and/or between intervention groups. These outcomes are intended to characterize intervention-associated alterations in gut microbiota composition.
Circulating adipokines assessed by serum analysis | Baseline, Week 12, and Week 20
  Adipokine profiling will be conducted on fasting serum samples collected at predefined study time points. Outcomes will include circulating concentrations of selected adipokines and the identification of adipokines showing significant changes between baseline and post-intervention time points and/or between intervention groups, reflecting alterations in adipose tissue-related endocrine function associated with the intervention.
Serum proteomic profile assessed by liquid chromatography-tandem mass spectrometry (LC-MS/MS) | Baseline, Week 12, and Week 20
  Proteomic profiling will be conducted on fasting serum samples collected at predefined study time points using LC-MS/MS. Primary proteomic outcomes will include relative protein abundances quantified based on normalized signal intensities and the identification of proteins showing significant differential expression between baseline and post-intervention time points and/or between intervention groups, reflecting molecular alterations associated with the intervention.
Serum metabolomic profile assessed by liquid chromatography-tandem mass spectrometry (LC-MS/MS) | Baseline, Week 12, and Week 20
  Metabolomic profiling will be conducted on fasting serum samples collected at predefined study time points using LC-MS/MS. Metabolomic outcomes will include relative abundances of detected metabolites quantified based on normalized signal intensities, as well as the identification of metabolites showing significant changes between baseline and post-intervention time points and/or between intervention groups, reflecting metabolic responses to the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Shan Gao, Doctoral degree, Study Chair — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to concerns regarding participant privacy and confidentiality, and because no formal plan for external data sharing has been established at this time.